CLINICAL TRIAL: NCT02040701
Title: Sleep Disordered Breathing in Children: Inflammation and Oxidative Stress
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: TASMC-13-RT-06-122-CTIL
Record Dates: First submitted 2014-01-09; First posted 2014-01-20 (Estimated); Last update posted 2014-01-20 (Estimated); Status verified 2014-01

CONDITIONS: Sleep Disordered Breathing (SDB); Endothelial Dysfunction
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 8 Weeks

GROUPS / COHORTS (2):
- SDB group
- Control group

SUMMARY:
The purpose of the study is to measure markers of inflammatory and oxidative stress known to be associated with cardiovascular morbidity in snoring children.

In addition, to measure markers of local inflammation and to evaluate the response to treatment.

ELIGIBILITY:
Inclusion Criteria:

* children ages 6 months-18 years
* suspected sleep-disordered breathing or will attend the pre-operative ENT clinic for adenoidectomy or adenotonsillectomy

Exclusion Criteria:

* craniofacial abnormalities
* neurological disorders
* genetic disorders
* infectious disease
* chronic inflammatory disease
* any underlying chronic medical condition

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: children ages 6 months-18 years who will undergo overnight sleep study at the Dana Children's hospital, Tel Aviv Medical Center because of snoring and suspected sleep-disordered breathing or will attend the pre-operative ENT clinic for adenoidectomy or adenotonsillectomy
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2006-05; Primary Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
Plasma inflammatory-markers | After the blood analyzed
  Sleep disordered breathing (SDB) in children is associated with increased markers of inflammation, atherogenesis and oxidative stress.

CONTACTS AND LOCATIONS:
Locations (1):
- Dana Children's hospital, Tel Aviv Medical Center, Tel Aviv, Israel